CLINICAL TRIAL: NCT02328066
Title: Diagnostic Accuracy of NICE Classification to Predict Deep Submucosal Invasion in Colon Lesions. Prospective Multicenter Study in Routine Clinical Practice
Brief Title: Diagnostic Accuracy of NICE Classification to Predict Deep Submucosal Invasion
Acronym: NICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asociación Española de Gastroenterología (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CEIC14/47
Record Dates: First submitted 2014-12-08; First posted 2014-12-31 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Colonic Polyps
Keywords: NBI; NICE classification; deep submucosal invasion; Colonic Polyps [C23.300.825.411.235]; Colonoscopy [E01.370.372.250.250.200]
MeSH Terms: conditions — Colonic Polyps | interventions — Narrow Band Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NBI used by trained endoscopists (Experimental): Assessment with NICE classification and NBI technology of colonic lesions (Paris classification type 0) greater than 1 cm found in a routine colonoscopy. This assessment was performed by previously trained endoscopists.
  Interventions: Device: NBI used by trained endoscopists

INTERVENTIONS:
Device: NBI used by trained endoscopists — Examination of colon lesions, using NBI and NICE classification, by endoscopists who previously performed an easy learning program. The learning program consists on the reading of two reference articles and a tutorial explaining the NICE classification. This tutorial shows several lesions and describes the characteristic features in which the classifications focus on.
  Other Names: Narrow Band Imaging; NICE classification

SUMMARY:
The purpose of this study is to evaluate the diagnostic accuracy of NICE classification to predict deep submucosal invasion of colonic polyps > 1 cm, considering histology as the gold standard, in a group of endoscopists who previously performed a training program.

DETAILED DESCRIPTION:
In the first phase of the study, a learning program of NICE classification based on examples will be performed. Forty images will be evaluated before and after the learning program.

In the second phase of the study, all consecutive patients who underwent to a colonoscopy will be included if a lesion greater than 1 cm is found and the endoscopy is performed with a high definition colonoscope with Narrow Band Imaging (NBI). Patients, lesions and endoscopy equipment characteristics will be recorded.

Subsequently, histological diagnosis of the lesion will also be recorded. Evaluated test (NICE classification) was blinded to the pathologist who performed the gold standard test (histology). In case of adenocarcinomas, histological predictors of lymph node metastases, with predefined assessment criteria, will also be recorded.

Finally, histological preparations of adenocarcinomas will be sent to the reference center and two experienced pathologists will examine them again.

ELIGIBILITY:
Inclusion patients criteria:

* Patients> 18 years
* Lesion Type 0 of Paris classification, greater than 1 cm, found in a colonoscopy performed by any medical indication with a high definition endoscope with Narrow Band Imaging.
* Achievable histology by endoscopic or surgical resection.
* Writing informed consent given.

Exclusion patients criteria:

* Age <18 years.
* Refusal to give informed consent.
* Contraindication for endoscopic or surgical resection.
* Urgent colonoscopy indication (eg severe rectorrhagia.).
* Patients with inflammatory bowel disease.
* Suspected metastatic neoplasia by previous imaging tests.

Exclusion lesions criteria:

* Polyp previously biopsied or resected.
* Poor preparation that does not allow a proper assessment of the lesion.
* NBI not performed.
* Unavailable or indefinite histology (endoscopic or surgical resection).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2171 (Actual)
Dates: Start 2014-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of NICE classification to predict deep submucosal invasion | 1 year
  Sensibility, specificity, negative predictive value and positive predictive value of NICE classification to predict deep submucosal invasion during routine colonoscopies.
  Gold standard (histology):
  * positive means adenocarcinoma with deep submucosal invasion (>1 mm)
  * negative means non adenocarcinoma or superficial adenocarcinoma (<1 mm)
  Evaluated test (NICE classification):
  * Positive means NICE type 3.
  * Negative means NICE type 1 and 2.
  Evaluated test (NICE classification) was blinded to the pathologist who performed the gold standard test (histology)

SECONDARY OUTCOMES:
Diagnostic accuracy of NICE classification to predict deep submucosal invasion in the pre-learning test | 0
  Sensibility, specificity, negative predictive value and positive predictive value of NICE classification to predict deep submucosal invasion in the pre-learning test.
Diagnostic accuracy of NICE classification to predict deep submucosal invasion in the post-learning test | 0
  Sensibility, specificity, negative predictive value and positive predictive value of NICE classification to predict deep submucosal invasion in the post-learning test (pre-clinical test)
Preplanned potential factors that could influence diagnostic accuracy of NICE classification | 1 year
  Related to the lesion: Size (mm); location: rectum/sigmoid/left colon/splenic flexure/transverse colon/hepatic flexure/right colon and cecum; Morphology according to the Paris classification (see categories in the reference article); Level of confidence: high/low; Successful complete submucosal injection: yes/no/not done; Chicken skin's sign: yes/no; Edges retraction: yes/no; Depressed areas: yes/no; Folds convergence: yes/no; Induration: yes/no; Obvious ulceration: yes/no; Polyp on polyp: yes/no; Technical resection: 8 categories according to the current practice.
  Related to the equipment: Colonoscope: 11 colonoscope models; Videoprocessor: Exera II, Exera III; Monitor: high definition, non-high definition
  Related to the endoscopist: Hospital type: Secondary or tertiary; Endoscopy experience (number of years); Previous experience in chromoendoscopy: yes/no; Previous experience in NBI: yes/no; Number of lesions included in the study; Review histology and images monthly: yes/no
Histological predictors of lymph node metastases of pT1 | 1 year
  * Histological type: adenocarcinoma, mucinous adenocarcinoma, cell carcinoma with signet ring, undifferentiated carcinoma, other.
  * Histologic Grade: Low Grade (well-moderately differentiated) or High-grade (poorly dif, undifferentiated, mucinous, signet ring).
  * Horizontal size of adenocarcinoma (mm)
  * Level of submucosal adenocarcinoma (mm)
  * Angiolymphatic invasion of small vessels: Present or absent
  * Perineural invasion: Present or Absent.
  * Tumor budding: Absent, Low grade (5-9 groups of 5 cells per field with 20x objective), High Grade (≥10 groups of 5 cells per field with 20x objective)
  * Polyp type that originated carcinoma: Tubular adenoma, Villous adenoma, Adenoma/sessile serrated polyp, Traditional serrated adenoma, Other
  * Resection margin: Negative or Positive
  * Size of negative margin (mm).

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Vega, Principal Investigator — Complexo Hospitalario de Ourense; Maria Luisa de Castro, Principal Investigator — Complexo Hospitalario Universitario de Vigo-CHUVI; Eva Martínez-Bauer, Principal Investigator — Corporacion Parc Tauli; Angel Fernández, Principal Investigator — Hospital Clínico de Zaragoza; Gema de la Poza, Principal Investigator — Hospital de Fuenlabrada; Jorge López, Principal Investigator — Hospital de Móstoles; Oscar Nogales, Principal Investigator — Gregorio Marañón Hospital; Beatriz Peñas, Principal Investigator — Hospital Universitario Ramon y Cajal; Pilar Díez, Principal Investigator — Hospital Río Ortega; Marta Hernández, Principal Investigator — Hospital Universitario Puerta de Hierro; Antonio Zebenzuy, Principal Investigator — Hospital Universitario de Canarias; Aurora Burgos, Principal Investigator — Hospital Universitario La Paz; Jorge Mendoza, Principal Investigator — Fundación de Investigación Biomédica - Hospital Universitario de La Princesa; Marco Antonio Álvarez, Principal Investigator — Hospital del Mar
Locations (1):
- Ignasi Puig, Manresa, Barcelona, Spain

REFERENCES:
- [Background] Hayashi N, Tanaka S, Hewett DG, Kaltenbach TR, Sano Y, Ponchon T, Saunders BP, Rex DK, Soetikno RM. Endoscopic prediction of deep submucosal invasive carcinoma: validation of the narrow-band imaging international colorectal endoscopic (NICE) classification. Gastrointest Endosc. 2013 Oct;78(4):625-32. doi: 10.1016/j.gie.2013.04.185. Epub 2013 Jul 30. PMID 23910062
- [Derived] Puig I, Lopez-Ceron M, Arnau A, Rosinol O, Cuatrecasas M, Herreros-de-Tejada A, Ferrandez A, Serra-Burriel M, Nogales O, Vida F, de Castro L, Lopez-Vicente J, Vega P, Alvarez-Gonzalez MA, Gonzalez-Santiago J, Hernandez-Conde M, Diez-Redondo P, Rivero-Sanchez L, Gimeno-Garcia AZ, Burgos A, Garcia-Alonso FJ, Bustamante-Balen M, Martinez-Bauer E, Penas B, Pellise M; EndoCAR group, Spanish Gastroenterological Association and the Spanish Digestive Endoscopy Society. Accuracy of the Narrow-Band Imaging International Colorectal Endoscopic Classification System in Identification of Deep Invasion in Colorectal Polyps. Gastroenterology. 2019 Jan;156(1):75-87. doi: 10.1053/j.gastro.2018.10.004. Epub 2018 Oct 6. PMID 30296432